CLINICAL TRIAL: NCT04962243
Title: Whether Patients With Achilles Tendon Tears Have Different Lipid Levels Than Healthy People: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019127
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing repair of Achilles tendon rupture: Patients undergoing repair of Achilles tendon rupture
  Interventions: Procedure: Repair surgery for Achilles tendon rupture
- Subjects who underwent physical examination during the same period: Subjects who underwent physical examination in the Physical Examination Center of Peking University Third Hospital during the same period

INTERVENTIONS:
Procedure: Repair surgery for Achilles tendon rupture — Repair surgery for Achilles tendon rupture
  Groups: Patients undergoing repair of Achilles tendon rupture

SUMMARY:
To explore the difference of blood lipid levels between patients with Achilles tendon rupture and healthy people without Achilles tendon rupture, and to provide clues for further exploration of its mechanism.

DETAILED DESCRIPTION:
Data were collected from 287 patients with Achilles tendon rupture repaired by Yang Yuping, deputy chief physician of the Institute of Sports Medicine of Peking University Third Hospital from January 2017 to December 2017. A total of 10,375 subjects who underwent physical examination in the Physical Examination Center of Peking University Third Hospital during the same period were selected as the control group, and 9,193 subjects were selected as the control group after excluding patients without blood lipid test results, professional athletes, hypertension and diabetes patients. The general data, blood glucose, blood lipid, blood uric acid, smoking and alcohol consumption of the subjects were collected through the hospital information system. The blood glucose, blood lipid, uric acid and other data of the control group and the Achilles tendon rupture group were detected, and it was concluded that the blood lipid level of the patients with Achilles tendon rupture group was higher than that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Rupture of Achilles tendon repair surgery experience

Exclusion Criteria:

* hypertension
* diabetes
* Professional athlete
* No blood lipid test results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Yang Yuping, Deputy Chief Physician of the Institute of Sports Medicine of Peking University Third Hospital from January 2017 to December 2017 in Peking University Third Hospital of Sports Medicine for patients with Achilles tendon rupture repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 10662 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | a month after the surgery
  Blood glucose levels of patients and control group were measured one month after surgery.
blood lipid levels | a month after the surgery
  blood lipid levels of patients and control group were measured one month after surgery.
uric acid levels | a month after the surgery
  uric acid levels of patients and control group were measured one month after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No